CLINICAL TRIAL: NCT05708053
Title: Cardio-protective Effect of Metformin in Patients Undergoing Elective Percutaneous Coronary Intervention
Brief Title: Cardio-protective Effect of Metformin in Patients Undergoing PCI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Future University in Egypt (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Radwa Abdelatif, Principal Investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: December-2019
Record Dates: First submitted 2023-01-09; First posted 2023-02-01 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Elective Percutaneous Coronary Intervention; Ischemic Reperfusion Injury
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin Group (Experimental): Patients will receive pre-treatment standard and post treatment of care to the procedure plus metformin 500 mg twice daily 7 days before and 6 months after the PCI procedure.
  Metformin will be stopped on the same day of the procedure and restored 3 hours after the procedure.
  Interventions: Drug: Metformin
- Comparator (No Intervention): Patients will receive pre-treatment and post treatment standard of care to the procedure

INTERVENTIONS:
Drug: Metformin — Metformin 500 mg twice
  Arms: Metformin Group

SUMMARY:
This is a two-arm randomized parallel study. Patients who will be meeting the above-mentioned criteria and agree to take part in the study, were asked to sign an informed consent prior conducting the study.

The whole study protocol were presented to the local institutional review board (IRB).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age above 18)
* Undergoing elective PCI

Exclusion Criteria:

1. Hypersensitivity to metformin or any component of the formulation
2. Patients with current or any history taking metformin either for diabetes mellitus or any other reason such as polycystic ovarian syndrome.
3. Patients diagnosed with type 1 or 2 diabetes mellitus.
4. Any oral or injectable hypoglycemic therapy (e.g. insulin, sulfonylureas)
5. Severe renal dysfunction (eGFR less than 30 mL/minute/1.73 m2 ) from any cause, including shock or septicemia; acute or chronic metabolic acidosis with or without coma (including diabetic ketoacidosis).
6. Treatment with systemic glucocorticoids within 3 months of randomization (due to its potential effect on plasma glucose and HbA1c levels).
7. Metabolic acidosis (total CO 2 below the laboratory lower limit of normal on most recent blood chemistry panel).
8. Need for coronary artery bypass grafting.
9. Participation in other clinical trial in the 30 days before enrollment.
10. The existence of a life-threatening disease with a life-expectancy of less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Postprocedural myocardial injury | 6 months
  the occurrence of postprocedural myocardial injury, defined as a postprocedural elevation of CKMB or cTnI more than 1 times the 99 th percentile of the URL [ 24 hours post PCI]

SECONDARY OUTCOMES:
CK-MB | 24 hours post PCI
  Mean peak values of CK-MB after intervention
cTn | 24 hours post PCI
  Mean peak values of cTnI after intervention
LVEF in percent | Baseline- 6 months
  Echo: to measure LVEF in percent
LVMI in g/m2 | Baseline- 6 months
  left ventricular mass index (LVMI) will be calculated in g/m2 using the sex and body surface area (m²) and measures of LVEDD in mm, IVSd in mm, PWd from the measures in the echocardiography
GFR | Baseline- monthly- 6 months
  glomerular filtration rate (GFR) will be calculated (unit ml/min) using age in years, sex, body weight in kilograms and serum creatinine in mg/dL
Serum creatinine (SCr) | Baseline- monthly- 6 months
  Serum creatinine (SCr) in mg/dL
Lactate concentration | Baseline - 6 months
  lactate concentration unit in mmol/L
Glucometabolic State | Baseline - 6 months
  Glucometabolic State using HbA1c (unit mmols/mol)
Incidence of Cardiovascular Event | Baseline - 6 months
  Cardiovascular events including major cardiac adverse events (MACE; death, recurrent MI, target lesion revascularization), stroke, non-elective hospitalizations for chest pain or heart failure, all recurrent coronary interventions, and internal cardiac defibrillator implantations. Mortality will be divided into cardiac and non- cardiac. Cardiac death will be divided into three categories: heart failure, sudden death, and others.
Rate of hospitalization | through study completion, an average of 6 months
  The number of hospitalizations within each group will be calculated during the study period.

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Faculty of Pharmacy, Cairo University, Cairo
  - Kasr El Aini Hospital, Cairo
  - Kasr El-Aini Hospital, Cairo

IPD SHARING:
Plan to Share IPD: Undecided